CLINICAL TRIAL: NCT03118687
Title: Human Immunome Program
Acronym: HIP
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Human Vaccines Project (Other)
Responsible Party: Principal Investigator, James E. Crowe, Jr., Principal Investigator, Vanderbilt University Medical Center
Other Study IDs: IRB#170398
Record Dates: First submitted 2017-04-13; First posted 2017-04-18 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Healthy
Keywords: Immune system

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Peripheral blood mononuclear cell (PBMCs)
  * Microbiome (stool, tongue, skin swabs)(optional)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Biospecimen and survey collection — Blood, microbiota, surveys/questionnaires, electronic medical records.

SUMMARY:
The Human Immunome Program is a large-scale, open-source effort seeking to fill a major gap in our knowledge of the immune system. The power of the immune system to fight disease lies in its ability recognize and adapt to an astonishing range of threats from viruses, parasites and bacteria to cancer cells. Underlying this ability is a vast but specific set of genes and molecular structures known as the human immunome, or the "parts list" of the immune system. This study aims to decipher the genetic sequences that make up this part list and link it to information about a person's microbiome composition and characteristics such as health history, race, and demographics over time. This information, made freely available to the public for use in research in de-identified form, will allow investigators to answer a wide variety of different questions about immune system function. This could transform how we diagnose, prevent and treat disease though the identification of new biomarkers while enabling highly targeted, computationally designed vaccines and therapies that reduce time and risk of product development.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female volunteers between the ages of 18 - 49 years of age at the time of first enrollment.
* Ability to comply: Participant willing and able to comply with the requirements of the protocol.
* Consent: Participants who have given informed consent for participation in the study

Exclusion Criteria:

Reason for exclusion throughout the entire study period:

* History of severe anemia requiring blood transfusion or current Hemoglobin < 10g/dL.
* Currently pregnant or pregnancy within 6 months.
* Current participation in another study resulting in blood collection which exceeds 550 ml in an 8 week period or occurs more frequently than 2 times per week.
* Temperature >101.4F
* Any condition which, in the opinion of the investigator, might interfere with study objectives.
* Any reason which, in the opinion of the investigator, adds additional risk to the patient.

Reason for exclusion in year 0 but not in year 1-9:

* History of known HIV infection or treatment.
* Immunosuppressive disease or use of systemic immunosuppressive therapy using drugs or cytotoxic agents including prednisone (IV, oral or inhaled) less than 6 months ago.
* History of diabetes mellitus -or a glucose (on CMP) ≥200 mg/dL.
* History of cancer including skin cancer.
* History of autoimmune disorders including but not limited to: Ulcerative colitis, Crohn's, Inflammatory Bowel Disease, Rheumatoid Arthritis, Scleroderma, Systemic lupus Erythematosus, Mixed Connective Tissue Disease, Graves, Autoimmune Thyroiditis, Hashimoto's Thyroiditis, Psoriasis, Multiple Sclerosis, Guillain-Barre Syndrome, Chronic Inflammatory demyelinating polyneuropathy, Myasthenia Gravis, Vasculitis, Alopecia areata, autoimmune hemolytic anemia, autoimmune hepatitis, dermatomyositis, idiopathic thrombocytopenic purpura, pemphigus, pernicious anemia, polyarteritis nodosa, polymyositis, Sjogren's Syndrome, Wegener's
* Severe obesity = (BMI >40 kg/m2).

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy adult volunteers
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2020-06-18 (Actual); Study Completion 2020-06-18 (Actual)

PRIMARY OUTCOMES:
The entire expressed B and T cell receptor repertoire ("Immunome") of the human immune system | 10 years
  The B and T cell receptor repertoire will be sequenced. The sequencing will continue until no new unique sequences appear.

CONTACTS AND LOCATIONS:
Overall Officials: James E Crowe Jr., M.D., Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- See also: The Human Vaccines Project is the parent project to the Human Immunome Program — http://humanvaccinesproject.org